CLINICAL TRIAL: NCT07095023
Title: A Single-Arm Clinical Study to Evaluate the Efficacy and Safety of Neoadjuvant Oral Paclitaxel Plus Fixed-Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Injection in Patients With HER2-positive Breast Cancer
Brief Title: Neoadjuvant Oral Paclitaxel Plus Subcutaneous Pertuzumab/Trastuzumab in Patients With HER2-positive Breast Cancer
Acronym: OPTIMAL-BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Peking University Shenzhen Hospital (Other); Hainan People's Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Nanfang Hospital, Southern Medical University (Other); Guangdong Women and Children Hospital (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Liu Qiang, Director, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-397-01
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancers
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Paclitaxel plus Subcutaneous Pertuzumab/Trastuzumab (Experimental): Paclitaxel oral solution plus subcutaneous fixed-dose combination of pertuzumab and trastuzumab
  Interventions: Drug: Paclitaxel oral solution plus Subcutaneous Pertuzumab/Trastuzumab

INTERVENTIONS:
Drug: Paclitaxel oral solution plus Subcutaneous Pertuzumab/Trastuzumab — Patients who meet the inclusion criteria will be enrolled and given paclitaxel oral solution and subcutaneous pertuzumab/trastuzumab for neoadjuvant treatment.
  Paclitaxel oral solution: 200mg/m2 po bid, D1,D8,D15, q3w. Subcutaneous pertuzumab/trastuzumab: 1200 mg pertuzumab plus 600 mg trastuzumab loading dose in 15 mL, followed by 600 mg pertuzumab plus 600 mg trastuzumab maintenance doses in 10 mL, q3w.
  Other Names: DHP107; RMX3001; Liporaxel; pertuzumab, trastuzumab, and hyaluronidase-zzxf

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of oral paclitaxel plus fixed-dose combination of pertuzumab and trastuzumab for subcutaneous injection in the neoadjuvant treatment of HER2+ breast cancer patients.

DETAILED DESCRIPTION:
OPTIMAL-BC is a multicenter, single arm study using a Simon's two-stage design evaluating neoadjuvant treatment with paclitaxel oral solution combined with subcutaneous fixed dose combination (FDC) of pertuzumab and trastuzumab every 3 weeks for 6 cycles. All subjects will undergo surgery in line with local guidelines following neoadjuvant therapy. The primary endpoint is total pathological complete response(tpCR, ypT0/is, ypN0).

ELIGIBILITY:
Inclusion Criteria:

Aged 18-70 years old. Histologically confirmed HER2-positive invasive breast cancer with clinical stages T1c-4, N0-3, and M0 (excluding T1cN0M0), according to the 8th American Joint Committee on Cancer (AJCC) edition BC staging system HER2 overexpression was defined as immunohistochemistry (IHC) 3+ or 2+ with HER2 gene amplification, determined by fluorescence in situ hybridization (FISH).

Baseline left ventricular ejection fraction (LVEF) of ≥50%. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.

The functional level of major organs must meet the following requirements (no blood transfusion and no use of white blood cell, red blood cell and platelet-raising drugs within 2 weeks before the first dose):

* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase and aspartate aminotransferase (ALT/AST) ≤1.5×ULN
* Blood urea nitrogen and serum creatinine ≤1.5×ULN
* Creatinine clearance (Ccr) ≥50 ml/min (Cockcroft-Gault formula) Signature of informed consent

Exclusion Criteria:

* History of invasive breast cancer. Bilateral breast cancer or inflammatory breast cancer . Prior excisional and/or incisional biopsy of the primary tumor and/or axillary lymph nodes.

Prior systemic therapy for breast cancer. History of life-threatening hypersensitivity reactions or known hypersensitivity to any component of the investigational drug.

Participation in another clinical trial of a drug or medical device within 4 weeks prior to the first dose and/or receipt of investigational drug/device during the trial.

Major surgery within 28 days prior to the first dose or planned major surgery during the study period.

History of other malignancies within the past 5 years, except for carcinoma in situ of the cervix, non-melanoma skin cancer, localized prostate cancer, or ductal carcinoma in situ.

Active tuberculosis or other severe infectious diseases requiring systemic treatment, including but not limited to bacteremia, severe pneumonia, and other serious infections.

History of immunodeficiency or autoimmune diseases, including but not limited to HIV infection (HIV antibody positive), systemic lupus erythematosus, rheumatoid arthritis, or history of organ transplantation.

History of cardiovascular or cerebrovascular diseases, including:

* Unstable angina;
* Clinically significant arrhythmias requiring medication;
* Myocardial infarction within the past 6 months;
* Heart failure or second-degree or higher atrioventricular block;
* Cerebral infarction (excluding lacunar infarction) or cerebral hemorrhage within the past 6 months.

Poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg despite regular medication), or history of hypertensive crisis or hypertensive encephalopathy.

Unsuitability for oral administration of the investigational drug, as judged by the investigator, including:

* Clinically significant or uncontrolled congenital or acquired gastrointestinal diseases;
* Diseases that may affect drug administration, gastric entry, or absorption (e.g., intestinal obstruction, Crohn's disease, ulcerative colitis).

Pregnant or breastfeeding women; women of childbearing potential with a positive pregnancy test at screening; or those unwilling to use effective contraception during the study and for 6 months after the last dose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Pathological Complete Response(tpCR) | Approximately 6 months from first dose of study drug following surgery or early withdrawal, whichever occurred first (Surgery was performed within 6 weeks after neoadjuvant treatment)
  It refers to the absence of any invasive cancer in the resected specimens (breast + axilla) after completion of neoadjuvant chemotherapy and surgery (i.e., ypT0/is, ypN0).

SECONDARY OUTCOMES:
Overall Response Rate(ORR) | Approximately 6 months from first dose of study drug following surgery or early withdrawal, whichever occurred first (Surgery was performed within 6 weeks after neoadjuvant treatment)
  Tumor assessments were made based upon the Response Evaluation Criteria in Solid Tumors (RECIST) criteria - version 1.1. ORR includes both partial response (PR) and complete response (CR).
Event-Free Survival (EFS) | Up to 3 years
  EFS is defined as the time from randomization to any of the following events: disease progression during neoadjuvant treatment, disease recurrence, or any cause of death.
Overall survival(OS) | Up to 3 years
  Overall survival is defined as the time from treatment start until death from any cause.
Health Related Quality of Life (QoL) | From baseline to 30 days after completion of treatment or the last follow-up visit
  To evaluate changes in health related quality of life (QoL) assessments from baseline in all subjects using the Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Scores in each dimension are uniformly transformed to dimensions ranging from 0 to 100. For functional and global quality of life scales, higher scores mean a better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms.
Adverse Events | From first dose of study drug to 30 days after completion of treatment
  Safety will be assessed by evaluating the incidence, and severity of adverse events according to CTCAE 5.0 (Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (9):
- China (9):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Guangdong Women and children Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Guangxi Provincial Cancer Hospital, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan Central Hospital, Haikou, Hainan
  - the First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University Shenzhen Hospita, Shenzhen

IPD SHARING:
Plan to Share IPD: No